CLINICAL TRIAL: NCT04801134
Title: Interventions to Manage Food Insecurity and Inappropriate Feeding Practices Related to the COVID-19 Pandemic (AMISTAD)
Brief Title: Interventions to Manage Food Insecurity and Inappropriate Feeding Practices Related to the COVID-19 Pandemic
Acronym: AMISTAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: Perrigo Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HRP-UT901
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Food Insecurity; Children, Only; Covid19
Keywords: Food Insecurity; COVID-19; Hispanic Children
MeSH Terms: conditions — COVID-19 | interventions — Educational Status; Community Resources

STUDY DESIGN:
Intervention Model Description: 50 families will be followed over 6 months, providing nutrition education and support with community resources to mitigate the families food insecurity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Food insecurity (Other): Food insecure families will be assigned education and community resources needed.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — as per previous description
  Other Names: Community Resources

SUMMARY:
This is a pilot study to determine how to identify and characterize effective approaches to assist Hispanic families who face food insecurity worsened by the Covid-19 pandemic. The investigators will enroll 50 children with food insecurity who are patients of the largest Federally Qualified Health Center in Austin, Texas. The investigators will follow them for 6 months, providing their caretakers with community resources, food literacy education and assisting them with web sites and applications that they can use to learn about and contact community assistance programs. The investigators will review food insecurity screening, qualitative interviews, dietary assessments, the child's anthropometrics, and standard of care laboratory results. The investigators will schedule follow up phone visits throughout the study to discuss with the families their needs and perceived assistance from the resources provided.

DETAILED DESCRIPTION:
The investigators propose to assess food insecurity and inappropriate feeding practices within a public health clinic patient population that has at least one child less than 2 years of age at home. A targeted intervention will determine whether focused family interactions with referral and follow-up to community agencies can mitigate the frequency and effects of food insecurity on children over a six-month period. Specifically, the investigators will identify 50 Hispanic families with food insecurity based on a full screen (the investigators expect to screen 150 families).

There are 2 in-person visits for this study, both of which are routine clinic visits where the child would be seen regardless of participation in this research study. The first visit at baseline will be when the subject is approached about the study and enrolled. The second visit will also be at a routine pediatric visit for medical care follow-up approximately 6 months later. Between in-person visits, phone calls for follow-up will take place.

The investigators will use a highly validated U.S. Department of Agriculture six-question, five-minute screening tool at each pediatric visit, via telehealth or in person. Those who screen as positive for food insecurity and consent to participate will be enrolled. Subjects will be enrolled as a parent/child dyad. The validated food-insecurity questionnaire will be completed at baseline, 3 months, and 6 months. The American Academy of Pediatrics recommends to screen for food insecurity as a standard of care.

Resources When appropriate, specific referrals will be made by the study personnel (PIs who are pediatricians) to food assistance programs including Good Apple, a local fresh produce delivery program, United Way of Central Texas, and local food banks. The participants will receive a call from the study coordinator who will review the family circumstances and plan for intervention with these partner programs and follow-up. A research team member will contact our food assistance partners to confirm each family's participation. The investigators will also confirm participation when available in WIC and SNAP programs. Partner organizations will provide financial data regarding the interventions they provide, which will be analyzed and interpreted within the context of families' participation in public programs such as WIC and SNAP. The study coordinator or designee who are part of the research study team will call the families frequently (weekly for first month, then every 2 weeks until 3 months, then monthly from 3-6 months; about 12-15 calls total) to check on their progress with the food assistance programs.

The participants will receive assistance with finding useful community resources websites and/or applications, grocery shopping lists, tips for shopping on a budget, and more topics related to nutrition, wellness, food assistance programs, food banks, bus routes, mindfulness, meal planning, and parenting strategies. Along with the referral resources, these documents and apps (i.e., My Fitness Pal food tracker, Pacer fitness tracker) will help the participants improve food literacy. Providing resources when a family is identified as food insecure is standard of care. However, the electronic resources and ongoing follow up are only related to this study. The investigators will track if the participants access the electronic resources that the investigators provide.

Education and Food Literacy Families will receive education about appropriate feeding practices with emphasis on not over-diluting infant formula and appropriate introduction of cow's milk, juice and solid foods.

Education for improving food literacy will focus on the following four dimensions from budgeting and planning, to food selection, to preparation and cooking, to eating.

Dietary Assessment Due to the relationship between dietary intake and overall health, dietary assessment tools are helpful to evaluate what a person is eating and how it may have an impact, either positive or negative, on their health. The participant will be asked to provide a 24-hour nutrition intake recall (describing types and amounts of foods and drinks they consumed the previous day) for themselves and their child. The study dietitian or designee will analyze the food records with nutrition software (i.e., NDSR) for macronutrient and macronutrient breakdown. Dietary intake will be assessed at baseline and after six months using a validated questionnaire. This information will be helpful to see how dietary intakes potentially change after enrollment and participation in community resources, and to see how dietary intakes affect growth in children.

Growth and Labs The investigators will compare growth measurements (weight, height or length, and head circumference) and dietary intakes of participating children at the start and after six months. In addition, the investigators will abstract data from the child's medical record for nutrition-related and routinely ordered labs (i.e., hemoglobin, lead level). These anthropometrics and laboratories are obtained as standard of care. Hemoglobin and lead levels usually are obtained at 1 and 2 years of age. Children screening out as iron deficient or with elevated lead levels will be managed by their pediatrician according to current American Academy of Pediatrics and Texas Department of Public Health guidelines.

Qualitative Interviews Qualitative interviews will be conducted in person or by phone at baseline and after three and six months to evaluate issues of concern such as child care, transportation and loss of employment. Qualitative interviews, pertaining to this study, will include asking participants which resources they found to be most useful, ease of navigating the resources, and their overall interactions with the partner organizations. All subjects will participate in the main (shorter) qualitative interview. Fifteen (15) subjects will be asked to participate in a longer qualitative interview, that the investigators expect to take an additional 30-60 minutes. These subjects will receive additional compensation for their time.

Standard of Care • Food insecurity screening, provision of referrals and resources to family, anthropometrics, labs, education

Research Activities

• Qualitative interviews, depression screen PHQ), anxiety screen (GAD), dietary assessment, follow-up with family to discuss their participation with referrals and resources

Our objectives are:

1. To identify and characterize Hispanic families who face food insecurity that occurred or worsened as a result of the current pandemic
2. To identify and characterize effective approaches to assisting families with inappropriate feeding practices, especially those related to infant formula preparation
3. To gain information regarding the types of resources that are most useful for planning purposes related to future pandemics or related public health crises
4. To define gaps in the process of obtaining and using available community resources
5. To provide baseline data regarding families and interventions so as to plan a larger-scale community-based assessment and intervention program

ELIGIBILITY:
Inclusion Criteria:

* Hispanic children, established patients of 2 participating CommUnityCare Clinics (FQHC) in Austin, TX, families that screened positive for food insecurity.

Exclusion Criteria:

* non-Hispanic children, families that screen negative for food insecurity, patients that do not receive medical care at the participating CommUnityCare clinics

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-03-22 (Estimated); Primary Completion 2022-03-22 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with mitigation of food insecurity as assessed by the "Six-item short form of the Household Food Security Scale", a validated 6 item food insecurity screening tool. | 6 months
  Mitigate food insecurity in participating families by providing education, community resources connections and close and frequent follow ups. Food insecurity will be assessed by the 6 item validated food insecurity screen periodically. The score is a sum of affirmative responses. Two or more affirmative responses indicate food insecurity; 5 or more affirmatives indicate hunger. (citation PMID 10432912)

SECONDARY OUTCOMES:
Types of community resources perceived as most helpful by the participants as assessed by a qualitative questionnaire. | 6 months
  Assess the benefits of various resources provided including electronic websites and applications, determining those resources that are most useful. This will be asked as an open question. Questionnaire is qualitative and therefore will not be scored.
Types of barriers to obtain assistance to alleviate food insecurity perceived by the participants as assessed by a qualitative questionnaire. | 6 months
  Identify any gaps or barriers in accessing the community resources. This will be asked as an open question. Questionnaire is qualitative and therefore will not be scored.

OTHER OUTCOMES:
Number of participants treated with intervention without evidence of impaired growth rate as measured in infantometer (length) and digital scale (weight). | 6 months
  length will be measured in centimeters in an infantometer with the child lying down without socks or shoes and weight will be measured in kilograms in a digital scale. Both measurements will be done by a medical assistant during each in-person visit to the clinic.
Number of participants treated with intervention with evidence of impaired growth rate | 6 months
  Growth rate data including Z-scores for height and weight will be measured at each family interaction. A decrease in a Z-score of > 0.25 (1/4 of a standard deviation) will be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Abrams, MD, Principal Investigator — University of Texas at Austin
Locations (1):
- CommUnityCare Health Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Patient information may be shared with the study sponsor and/or representative of the sponsor; representatives of UT Austin and the UT Austin Institutional Review Board; Other collaborating organizations (Good Apple, United Way of Central Texas, local food banks, WIC, SNAP). However, we will not share the subjects' data or samples with other researchers for future research studies.

REFERENCES:
- [Background] Blumberg SJ, Bialostosky K, Hamilton WL, Briefel RR. The effectiveness of a short form of the Household Food Security Scale. Am J Public Health. 1999 Aug;89(8):1231-4. doi: 10.2105/ajph.89.8.1231. PMID 10432912
- [Result] Shi Q, Castillo F, Viswanathan K, Kupferman F, MacDermid JC. Facilitators and Barriers to Access to Pediatric Medical Services in a Community Hospital. J Prim Care Community Health. 2020 Jan-Dec;11:2150132720904518. doi: 10.1177/2150132720904518. PMID 31997703
- [Result] Peltz A, Garg A. Food Insecurity and Health Care Use. Pediatrics. 2019 Oct;144(4):e20190347. doi: 10.1542/peds.2019-0347. Epub 2019 Sep 9. PMID 31501238
- [Result] COUNCIL ON COMMUNITY PEDIATRICS; COMMITTEE ON NUTRITION. Promoting Food Security for All Children. Pediatrics. 2015 Nov;136(5):e1431-8. doi: 10.1542/peds.2015-3301. PMID 26498462
- [Result] Nicola M, Alsafi Z, Sohrabi C, Kerwan A, Al-Jabir A, Iosifidis C, Agha M, Agha R. The socio-economic implications of the coronavirus pandemic (COVID-19): A review. Int J Surg. 2020 Jun;78:185-193. doi: 10.1016/j.ijsu.2020.04.018. Epub 2020 Apr 17. PMID 32305533
- [Result] Keenan DP, Olson C, Hersey JC, Parmer SM. Measures of food insecurity/security. J Nutr Educ. 2001;33 Suppl 1:S49-58. doi: 10.1016/s1499-4046(06)60069-9. PMID 12857544
- [Result] Kaiser LL, Melgar-Quinonez H, Townsend MS, Nicholson Y, Fujii ML, Martin AC, Lamp CL. Food insecurity and food supplies in Latino households with young children. J Nutr Educ Behav. 2003 May-Jun;35(3):148-53. doi: 10.1016/s1499-4046(06)60199-1. PMID 12773286
- [Result] Matheson DM, Varady J, Varady A, Killen JD. Household food security and nutritional status of Hispanic children in the fifth grade. Am J Clin Nutr. 2002 Jul;76(1):210-7. doi: 10.1093/ajcn/76.1.210. PMID 12081837
- See also: Map the Meal Gap is an annual study designed to improve the understanding of food insecurity and food costs at a local level — https://map.feedingamerica.org/county/2017/overall/texas/county/travis
- See also: information on food and nutrition assistance program/USDA — http://www.fns.usda.gov/